CLINICAL TRIAL: NCT00303108
Title: Phase II Study of Doxil and Carboplatin, Plus Herceptin in HER2+ Patients, in Metastatic Breast Cancer
Brief Title: Doxil & Carboplatin Plus HER2+ in Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: US Oncology Research (Industry)
Collaborators: Ortho Biotech, Inc. (Industry); Tibotec Pharmaceutical Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 04111
Record Dates: First submitted 2006-03-13; First posted 2006-03-15 (Estimated); Results first posted 2016-11-03 (Estimated); Last update posted 2016-11-03 (Estimated); Status verified 2016-09

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — liposomal doxorubicin; Carboplatin; Trastuzumab

ARMS (1):
- Arm 1 (Experimental): Patients will receive IV Doxil 30 mg/m2 and carboplatin AUC=5 on Day 1 of each cycle. A cycle consists of 28 days. In addition, HER2+ (IHC3+ and FISH+) patients only will receive a one-time loading dose of Herceptin 8 mg/kg IV on Day 1 of Cycle 1 and 4 mg/kg on Day 1 and Day 15 of every cycle thereafter.
  Interventions: Drug: Pegylated liposomal doxorubicin; Drug: Carboplatin; Drug: trastuzumab

INTERVENTIONS:
Drug: Pegylated liposomal doxorubicin — 30 mg/m2 IV on Day 1 of each 28 day cycle
  Other Names: Doxil
Drug: Carboplatin — AUC=5 on Day 1 of each 28 day cycle
Drug: trastuzumab — 4 mg/kg on Days 1 and 15 of each cycle(loading dose of 8 mg/kg on Day 1 of Cycle 1 only)
  Other Names: Herceptin

SUMMARY:
The purpose of this study is to determine the ORR associated with Doxil in combination with carboplatin in HER2- (negative) MBC (and with Herceptin in HER2+ MBC).

ELIGIBILITY:
Inclusion Criteria:

* Has metastatic breast cancer with documented HER2- or HER2+ (IHC3+ or FISH+) disease
* Has measurable MBC, with at least 1 measurable lesion per RECIST criteria (see Section 10). Irradiated lesions cannot be used to assess response but can be used to assess progression.
* Has had no prior treatment with Doxil or carboplatin; may have had adjuvant Herceptin if treatment was completed more than 1 year prior to study
* Has had no adjuvant chemotherapy within 1 year prior to study, but may have received prior anthracyclines as adjuvant chemotherapy
* For taxane-pretreated patients (adjuvant or metastatic), has had no more than 1 prior chemotherapy regimen for MBC
* For taxane-naïve patients, has had no prior chemotherapy for MBC
* Has had cumulative doses of < 300 mg/m2 prior doxorubicin or < 450 mg/m2 prior epirubicin
* Has normal cardiac function as evidenced by a LVEF within institutional normal limits by multiple gated acquisition (MUGA) scan. An echocardiogram (ECHO) may be used if MUGA is not available, but the same test must be used throughout the study to evaluate LVEF.
* Has an ECOG Performance Status (PS) 0-2 (see Appendix I)
* Is a male or female greater than or equal to 18 years of age
* Laboratory Values - Please refer to protocol section 4.2 for specific laboratory values.
* Has a negative serum pregnancy test within 7 days prior to registration (woman of childbearing potential [WOCBP; not surgically sterilized and between menarche and 1 year postmenopause])
* If fertile, patient (male or female) has agreed to use an acceptable method of birth control (eg, abstinence, intrauterine device, oral contraceptives, barrier device with spermicide or surgical sterilization) to avoid pregnancy for the duration of the study and for a period of 3 months thereafter.
* Has signed a Patient Informed Consent Form
* Has signed a Patient Authorization Form (HIPAA Form)
* Has a life expectancy of > 3 months

Exclusion Criteria:

* Has had a myocardial infarction (MI) within 6 months of trial enrollment, or has New York Heart Association (NYHA; see Appendix IV) Class II or greater heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, clinically significant pericardial disease, or electrocardiographic evidence of acute ischemic or active conduction system abnormalities
* Has a history of hypersensitivity reactions attributed to a conventional formulation of doxorubicin HCL or the components of Doxil
* Has evaluable only disease; eg, bone only, pleural, peritoneal only disease
* Is receiving concurrent immunotherapy, hormonal therapy, or radiation therapy. Patients receiving immunosuppressant therapy for autoimmune disease may enroll on the trial after a drug washout period of 2 weeks.
* Is receiving concurrent investigational therapy or has received such therapy within 30 days
* Has evidence of brain metastases requiring steroids and/or radiation or any documented leptomeningeal disease
* Has a serious uncontrolled intercurrent medical or psychiatric illness, including serious infection or history of uncontrolled seizures, CNS disorders deemed by the Treating Physician to be clinically significant, precluding informed consent
* Has a history of other malignancy within the last 5 years (except cured basal cell carcinoma of skin and carcinoma in situ of uterine cervix), which could affect the diagnosis or assessment of any of the study drugs
* Is a pregnant or lactating woman
* Is unable to comply with requirements of study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2005-12; Primary Completion 2010-03 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rufus P Collea, MD, Principal Investigator — US Oncology Research
Locations (56):
- United States (56):
  - Birmingham Hematology and Oncology, Birmingham, Alabama
  - Hematology Oncology Associates, Phoenix, Arizona
  - Northern AZ Hematology & Oncology Associates-Sedona, Sedona, Arizona
  - Rocky Mountain Cancer Center-Rose, Denver, Colorado
  - Florida Cancer Institute, New Port Richey, Florida
  - Ocala Oncology Center, Ocala, Florida
  - Hematology Oncology Associates of IL, Chicago, Illinois
  - Cancer Care & Hematology Specialists of Chicagoland, PC, Niles, Illinois
  - Central Indiana Cancer Centers, Indianapolis, Indiana
  - Kansas City Cancer Centers-Southwest, Overland Park, Kansas
  - Maryland Oncology Hematology, PA, Columbia, Maryland
  - Flavio Kruter, MD, PA, Westminster, Maryland
  - Minnesota Oncology Hematology, PA, Minneapolis, Minnesota
  - Missouri Cancer Associates, Columbia, Missouri
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - New Mexico Cancer Care Associates, Santa Fe, New Mexico
  - New York Oncology Hematology, PC, Albany, New York
  - Ruth Oratz MD, New York, New York
  - Raleigh Hematology Oncology Associates, Cary, North Carolina
  - Greater Dayton Cancer Center, Kettering, Ohio
  - Willamette Vallejy Cancer Center, Eugene, Oregon
  - Medical Oncology Associates, Kingston, Pennsylvania
  - Texas Cancer Center - Abilene (South), Abilene, Texas
  - Texas Oncology, P.A.-Amarillo, Amarillo, Texas
  - Texas Cancer Center, Arlington, Texas
  - Mamie McFaddin Ward Cancer Center, Beaumont, Texas
  - Texas Oncology, PA-Bedford, Bedford, Texas
  - Texas Cancer Center at Medical City, Dallas, Texas
  - Texas Oncology, PA, Dallas, Texas
  - The TexasCancer Center, Dallas, Texas
  - Texas Cancer Center-Denton, Denton, Texas
  - El Paso Cancer Treatment Ctr, El Paso, Texas
  - Texas Oncology, PA, Fort Worth, Texas
  - Texas Oncology, PA, Garland, Texas
  - Texas Oncology, PA, Houston, Texas
  - Lake Vista Cancer Center, Lewisville, Texas
  - Longview Cancer Center, Longview, Texas
  - South Texas Cancer Center-McAllen, McAllen, Texas
  - Texas Cancer Center of Mesquite, Mesquite, Texas
  - Alison Cancer Center, Midland, Texas
  - West Texas Cancer Center, Odessa, Texas
  - Paris Regional Cancer Center, Paris, Texas
  - HOAST-Medical Dr., San Antonio, Texas
  - Texas Cancer Center-Sherman, Sherman, Texas
  - Texas Oncology Cancer Center-Sugar Land, Sugar Land, Texas
  - Tyler Cancer Center, Tyler, Texas
  - Texas Oncology Cancer Care and Research Center-Waco, Waco, Texas
  - Texas Oncology, P.A., Webster, Texas
  - Fairfax Northern VA Hem-Onc PC, Fairfax, Virginia
  - Virginia Oncology Associates, Norfolk, Virginia
  - Onc and Hem Associates of SW VA, Inc, Salem, Virginia
  - Puget Sound Cancer Center-Edmonds, Edmonds, Washington
  - Puget Sound Cancer Center-Seattle, Seattle, Washington
  - Cancer Care Northwest-North, Spokane, Washington
  - Northwest Cancer Specialists-Vancouver, Vancouver, Washington
  - Yakima Valley Mem Hosp/North Star Lodge, Yakima, Washington

REFERENCES:
- [Derived] Collea RP, Kruter FW, Cantrell JE, George TK, Kruger S, Favret AM, Lindquist DL, Melnyk AM, Pluenneke RE, Shao SH, Crockett MW, Asmar L, O'Shaughnessy J. Pegylated liposomal doxorubicin plus carboplatin in patients with metastatic breast cancer: a phase II study. Ann Oncol. 2012 Oct;23(10):2599-2605. doi: 10.1093/annonc/mds052. Epub 2012 Mar 19. PMID 22431702

RESULTS

PARTICIPANT FLOW:
Groups:
- D+C and Taxane Naive: Doxil, Carboplatin and Taxane naive
- D+C and Taxane Pretreated: Doxil, Carboplatin and Taxane pretreated
- D+C+H: Doxil, Carboplatin, and Herceptin
Period: Overall Study
Arm/Group | D+C and Taxane Naive | D+C and Taxane Pretreated | D+C+H
Started | 43 | 46 | 47
Completed | 31 | 37 | 31
Not Completed | 12 | 9 | 16
Not completed — Adverse Event | 5 | 6 | 7
Not completed — Patient Request | 4 | 2 | 8
Not completed — Failed Entry | 1 | 0 | 1
Not completed — ineligible | 2 | 1 | 0

BASELINE CHARACTERISTICS:
Population: ITT population
Groups:
- Total: Total of all reporting groups
Arm/Group | D+C and Taxane Naive | D+C and Taxane Pretreated | D+C+H | Total
Number analyzed (Participants) | 43 | 46 | 47 | 136
Age, Continuous [Median (Full Range); unit: years] | 61.0 [28.0 to 84.9] | 51.7 [29.8 to 72.3] | 54.1 [29.0 to 77.6] | 56.4 [28.0 to 84.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 46 | 47 | 135
  Male | 1 | 0 | 0 | 1
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 30 | 34 | 37 | 101
  Black | 10 | 8 | 7 | 25
  Hispanic | 3 | 4 | 2 | 9
  Hawaiian | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 43 | 46 | 47 | 136

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Objective response (OR) = CR + PR.
Time Frame: From date of randomization until the date of first documented progression or date of intolerable toxicity, whichever came first, assessed up to 54 months.
Population: Evaluable population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | D+C and Taxane Naive | D+C and Taxane Pretreated | D+C+H
Number analyzed (Participants) | 39 | 42 | 45
percentage of participants | 30.8 [17.0 to 47.6] | 31.0 [17.6 to 47.1] | 55.6 [40.0 to 70.4]

2. Secondary Outcome: Duration of Response
Description: Duration from date of stating treatment to the date of first CR or PR.
Time Frame: as for outcome 1
Population: Patients who achieved CR or PR.
Measure: Median (Full Range); unit: months
Arm/Group | D+C and Taxane Naive | D+C and Taxane Pretreated | D+C+H
Number analyzed (Participants) | 12 | 13 | 25
months | 11.1 [0.9 to 15.2] | 7.0 [2.8 to 13.2] | 11.8 [2.3 to 16.8]

3. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS is measured from the date of randomization to the date of first documented disease progression or date of death, whichever comes first. If a patient neither progresses nor dies, this patient will be censored at last contact date.
  Progression is defined as appearance of one or more new lesions. Unequivocal progression of existing non-target lesions. Although a clear progression of "non-target" lesions only is exceptional, in such circumstances, the opinion of the Treating Physician should prevail, and the progression status should be confirmed at a later time by the review panel.
Time Frame: 30 months
Population: ITT population
Measure: Median (Full Range); unit: months
Arm/Group | D+C and Taxane Naive | D+C and Taxane Pretreated | D+C+H
Number analyzed (Participants) | 43 | 46 | 47
months | 8.1 [0.3 to 28.5] | 5.4 [0.1 to 21.0] | 10.1 [0.2 to 18.5]

4. Secondary Outcome: 1-year Overall Survival
Description: OS is measured from the date of randomization to the date of death for a dead patient. If a patient is still alive or is lost to follow up, the patient will be censored at the last contact date.
Time Frame: 1 year
Population: ITT population
Measure: Number (95% Confidence Interval); unit: probability of overall survival
Arm/Group | D+C and Taxane Naive | D+C and Taxane Pretreated | D+C+H
Number analyzed (Participants) | 43 | 46 | 47
probability of overall survival | 0.83 [0.67 to 0.915] | 0.56 [0.40 to 0.69] | 0.90 [0.76 to 0.96]

ADVERSE EVENTS:
Time Frame: During the whole treatment period, up to 30 days following last dose.
Groups:
- D+C and Taxane Naive or Pretreated: Doxil, Carboplatin and Taxane naive or pretreated.
Arm/Group | D+C and Taxane Naive or Pretreated | D+C+H
Serious Adverse Events (participants affected / at risk) | 8/83 | 3/46
Other Adverse Events (participants affected / at risk) | 80/83 | 44/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | D+C and Taxane Naive or Pretreated (N=83) | D+C+H (N=46)
ANEMIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
ANOREXIA (Gastrointestinal disorders) | 1 (1) | 0 (0)
DEHYDRATION (Gastrointestinal disorders) | 2 (3) | 0 (0)
NAUSEA AND VOMITING (Gastrointestinal disorders) | 0 (0) | 2 (2)
PANCYTOPENIA (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
PNEUMONIA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
RENAL FAILURE ACUTE (Renal and urinary disorders) | 1 (1) | 0 (0)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
URINARY TRACT INFECTION (Renal and urinary disorders) | 1 (1) | 0 (0)
VOMITING (Gastrointestinal disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | D+C and Taxane Naive or Pretreated (N=83) | D+C+H (N=46)
ALLERGIC REACTION (Immune system disorders) | 5 (6) | 2 (2)
ALOPECIA (Skin and subcutaneous tissue disorders) | 11 (11) | 15 (17)
ANEMIA (Blood and lymphatic system disorders) | 48 (152) | 30 (90)
ANOREXIA (Gastrointestinal disorders) | 12 (14) | 11 (11)
CONSTIPATION (Gastrointestinal disorders) | 20 (24) | 8 (8)
DEHYDRATION (Gastrointestinal disorders) | 1 (1) | 3 (3)
DIARRHEA (Gastrointestinal disorders) | 12 (16) | 9 (15)
DIZZINESS (Nervous system disorders) | 5 (7) | 1 (1)
DRY SKIN (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (4)
DYSPEPSIA (Gastrointestinal disorders) | 1 (1) | 3 (3)
EDEMA (Blood and lymphatic system disorders) | 7 (7) | 4 (11)
FEVER (General disorders) | 3 (3) | 4 (5)
FLUSHING (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
HAND-FOOT SYNDROME (Skin and subcutaneous tissue disorders) | 8 (15) | 7 (10)
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 1 (2) | 4 (7)
HYPOKALEMIA (Metabolism and nutrition disorders) | 1 (4) | 3 (3)
INSOMNIA (General disorders) | 6 (6) | 3 (3)
LEUCOPENIA (Blood and lymphatic system disorders) | 21 (64) | 18 (75)
MUCOSITIS (Infections and infestations) | 6 (11) | 10 (20)
MUSCLE WEAKNESS (Musculoskeletal and connective tissue disorders) | 6 (8) | 3 (5)
MYALGIA (Musculoskeletal and connective tissue disorders) | 3 (4) | 6 (6)
NAIL DISORDER (Skin and subcutaneous tissue disorders) | 2 (2) | 4 (6)
NAUSEA (Gastrointestinal disorders) | 43 (88) | 29 (44)
NEUROPATHY (Nervous system disorders) | 4 (4) | 4 (5)
NEUTROPENIA (Blood and lymphatic system disorders) | 40 (177) | 26 (145)
PAIN BONE (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (5)
RASH (Skin and subcutaneous tissue disorders) | 8 (10) | 9 (15)
SHORTNESS OF BREATH (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 4 (4)
STOMATITIS (Gastrointestinal disorders) | 5 (7) | 1 (1)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 35 (139) | 14 (82)
VOMITING (Gastrointestinal disorders) | 16 (27) | 12 (14)
WEAKNESS (General disorders) | 40 (85) | 23 (41)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No